CLINICAL TRIAL: NCT06865625
Title: The Effect of Using a Smart Phone App on Oral Hygiene and Brushing Training During Fixed Orthodontic Therapy
Brief Title: Smartphone App Impact on Oral Hygiene in Orthodontics
Status: Completed | Type: Observational
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Seda Sağoğlu, Principal Investigator / Research Assistant, Konya Necmettin Erbakan Üniversitesi
Other Study IDs: 2023/319
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Oral Hygiene Education Methods
Keywords: mobile application

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Dentabuddy Group with good oral hygiene: Individuals with good oral hygiene receiving oral hygiene education through the Dentabuddy application.
  Interventions: Behavioral: mobile application
- Dentabuddy Group with fair oral hygiene: Individuals with fair oral hygiene receiving oral hygiene education through the Dentabuddy application.
  Interventions: Behavioral: mobile application
- Dentabuddy Group with poor oral hygiene: Individuals with poor oral hygiene receiving oral hygiene education through the Dentabuddy application.
  Interventions: Behavioral: mobile application
- Assistant based trainning with good oral hygiene Group: Individuals with good oral hygiene receiving oral hygiene education through traditional methods.
  Interventions: Behavioral: traditional oral hygiene motivation
- Assistant based trainning with fair oral hygiene Group: Individuals with fair oral hygiene receiving oral hygiene education through traditional methods.
  Interventions: Behavioral: traditional oral hygiene motivation
- Assistant based trainning with poor oral hygiene Group: Individuals with poor oral hygiene receiving oral hygiene education through traditional methods.
  Interventions: Behavioral: traditional oral hygiene motivation

INTERVENTIONS:
Behavioral: mobile application — In this study, unlike similar studies in the literature, participants were grouped based on their oral hygiene status.
  Groups: Dentabuddy Group with fair oral hygiene; Dentabuddy Group with good oral hygiene; Dentabuddy Group with poor oral hygiene
Behavioral: traditional oral hygiene motivation — The group demonstrating the brushing technique on a braces model
  Groups: Assistant based trainning with fair oral hygiene Group; Assistant based trainning with good oral hygiene Group; Assistant based trainning with poor oral hygiene Group

SUMMARY:
This study aimed to compare changes in gingival index (GI), plaque index (PI), and gingival bleeding index (GBI) values in fixed orthodontic patients. Participants were classified into two groups based on their oral hygiene: those using the Dentabuddy app for oral hygiene improvement and those receiving assistant-led toothbrushing training.

Will the use of the Dentabuddy application lead to differences in oral hygiene levels? Can adolescents effectively utilize the program? Participants will compare the effectiveness of the smartphone application with a group receiving traditional oral hygiene motivation.

Participants:

Will use the program according to the designated time intervals. Will attend their appointments regularly.

DETAILED DESCRIPTION:
The Dentabuddy application is a free oral hygiene improvement tool available for download on the Google Play Store. This study will include 60 patients aged 12-18 years who have been undergoing fixed orthodontic treatment for at least six months. Patients will be classified into good, fair, and poor oral hygiene groups based on the Simplified Oral Hygiene Index (OHI-S), assessed by the second researcher. Using the Research Randomizer website, participants will be randomly assigned to either the Dentabuddy group or the assistant-supported training group.

Gingival Index (GI), Plaque Index (PI), and Gingival Bleeding Index (GBI) values will be recorded at baseline, after one month, and after three months. These data will be compared between groups. Additionally, at the end of three months, participants will be asked to demonstrate the brushing technique they were taught using a bracketed model. Those meeting specific criteria will be classified as having successfully demonstrated the brushing technique.

ELIGIBILITY:
Inclusion Criteria:

* no missing teeth,
* no systemic diseases or medications,
* complete permanent dentition,
* ability to maintain personal oral hygiene

Exclusion Criteria:

* dental treatment affecting oral hygiene

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Faculty of Dentistry
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Oral hygiene in patients undergoing fixed orthodontic treatment | From August to November 2023
  Participants whose oral hygiene scores are monitored through the use of the Dentabuddy application.
  The Gingival Index (GI) and Plaque Index (PI) are assessed on four surfaces of each tooth (mesial, distal, buccal/labial, and lingual) using a scale from 0 to 3. The total score from all evaluated sites is summed and divided by the total number of teeth to obtain the mean GI and PI values. A reduction in values will indicate a positive outcome of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Sağoğlu, Research Assistant, Principal Investigator — Konya Necmettin Erbaka University Faculty of Dentistry
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zotti F, Dalessandri D, Salgarello S, Piancino M, Bonetti S, Visconti L, Paganelli C. Usefulness of an app in improving oral hygiene compliance in adolescent orthodontic patients. Angle Orthod. 2016 Jan;86(1):101-7. doi: 10.2319/010915-19.1. Epub 2015 Mar 23. PMID 25799001